CLINICAL TRIAL: NCT01371838
Title: A Phase III, Multicentre, Randomised, Double-Blind, Comparative Study to Evaluate the Efficacy and Safety of Intravenous Ceftaroline Versus Intravenous Ceftriaxone in the Treatment of Adult Hospitalised Patients With Community-Acquired Bacterial Pneumonia in Asia
Brief Title: A Study to Evaluate the Efficacy and Safety of Intravenous Ceftaroline Versus Intravenous Ceftriaxone in the Treatment of Adult Hospitalised Patients With Community-Acquired Bacterial Pneumonia in Asia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3720C00002
Record Dates: First submitted 2011-04-27; First posted 2011-06-13 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Community-Acquired Bacterial Pneumonia; Lung Infection of Individual Not Recently Hospitalized
Keywords: Community-Acquired Bacterial Pneumonia
MeSH Terms: interventions — Ceftaroline; Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Ceftaroline (Experimental)
  Interventions: Drug: Ceftaroline
- Ceftriaxone plus placebo (Active Comparator)
  Interventions: Drug: Ceftriaxone

INTERVENTIONS:
Drug: Ceftaroline — Two consecutive infusions q12h for 5 to 7 days
  Arms: Ceftaroline
Drug: Ceftriaxone — One dose infusion followed by IV saline placebo infused q24h for 5 to 7 days plus two consecutive saline placebo infusion q24h.
  Arms: Ceftriaxone plus placebo

SUMMARY:
This purpose of this study is to Evaluate the Efficacy and Safety of Intravenous Ceftaroline Versus Intravenous Ceftriaxone in the Treatment of Adult Hospitalised Patients With Community-Acquired Bacterial Pneumonia in Asia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 or more years of age
* Lung Infection of Individual not Recently Hospitalized meeting the following criteria: Radiographically-confirmed pneumonia (new or progressive infection site of the lungs) consistent with bacterial pneumonia), AND Acute illness (≤ 7 days duration) with at least three of the following clinical signs or symptoms consistent with lung infection: New or increased cough, Purulent sputum or change in sputum character, Auscultatory findings consistent with pneumonia, Difficulty in breathing, short breath, or decreased partial pressure of oxygen in blood, Fever greater than 38ºC oral or body temperature lower than that required for normal body function(< 35ºC), White blood cell count greater than or less than the normal, Greater than 15% immature neutrophils (bands) irrespective of white blood cell count, AND Moderate lung infection
* The subject must require initial hospitalization, or treatment in an emergency room or urgent care setting, by the standard of care
* The subject's infection would require initial treatment with intravenous antimicrobials
* Female subjects of child-bearing potential, and those who are fewer than 2 years post-menopausal, must agree to, and comply with, using highly effective methods of birth control while participating in this study

Exclusion Criteria:

* Lung Infection of Individual not Recently Hospitalized suitable for outpatient therapy with an oral antimicrobial agent
* Confirmed or suspected respiratory tract infections attributable to sources other than bacteria from the individuals not recently hospitalized(e.g., ventilator-associated pneumonia, hospital-acquired pneumonia, visible/gross aspiration pneumonia, suspected viral, fungal, or mycobacterial infection of the lung)
* Non-infectious causes of lung lesion (e.g., pulmonary embolism, chemical pneumonitis from aspiration, hypersensitivity pneumonia, congestive heart failure)
* Accumulation of pus in the pleural cavity
* Microbiologically-documented infection with a pathogen known to be resistant to ceftriaxone, or epidemiological or clinical context suggesting high likelihood of a ceftriaxone-resistant "typical" bacterial pathogen.

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 848 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, Study Director — AstraZeneca
Locations (43):
- China (13):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jiangyin
  - Research Site, Nanchang
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Wuxi
- India (12):
  - Research Site, Bangalore
  - Research Site, Calicut
  - Research Site, Goa
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Lucknow
  - Research Site, Ludhiana
  - Research Site, Mysore
  - Research Site, New Delhi
  - Research Site, Trivandrum
  - Research Site, Varanasi
  - Research Site, Vellore
- South Korea (10):
  - Research Site, Anyang-si
  - Research Site, Bucheon-si
  - Research Site, Cheonan-si
  - Research Site, Chuncheon
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Wŏnju
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, Taichung
  - Research Site, Taipei
- Vietnam (4):
  - Research Site, Can Tho
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

REFERENCES:
- [Derived] Zhuo C, Huang Y, Liu W, Xu JF, Zhu WY, Stone GG, Yan JL, Mohamed N. Efficacy and Safety of Ceftaroline Fosamil in Hospitalized Patients with Community-Acquired Pneumonia in China: Subset Analysis of an International Phase 3 Randomized Controlled Trial. Infect Drug Resist. 2022 Feb 23;15:605-617. doi: 10.2147/IDR.S342558. eCollection 2022. PMID 35237053
- [Derived] Dryden M, Kantecki M, Yan JL, Stone GG, Leister-Tebbe H, Wilcox M. Treatment outcomes of secondary bacteraemia in patients treated with ceftaroline fosamil: pooled results from six phase III clinical trials. J Glob Antimicrob Resist. 2022 Mar;28:108-114. doi: 10.1016/j.jgar.2021.10.027. Epub 2021 Dec 16. PMID 34922058
- [Derived] Li J, Das S, Zhou D, Al-Huniti N. Population Pharmacokinetic Modeling and Probability of Target Attainment Analyses in Asian Patients With Community-Acquired Pneumonia Treated With Ceftaroline Fosamil. Clin Pharmacol Drug Dev. 2019 Jul;8(5):682-694. doi: 10.1002/cpdd.673. Epub 2019 May 1. PMID 31044546
- [Derived] Cheng K, Pypstra R, Yan JL, Hammond J. Summary of the safety and tolerability of two treatment regimens of ceftaroline fosamil: 600 mg every 8 h versus 600 mg every 12 h. J Antimicrob Chemother. 2019 Apr 1;74(4):1086-1091. doi: 10.1093/jac/dky519. PMID 30597021
- [Derived] Das S, Li J, Iaconis J, Zhou D, Stone GG, Yan JL, Melnick D. Ceftaroline fosamil doses and breakpoints for Staphylococcus aureus in complicated skin and soft tissue infections. J Antimicrob Chemother. 2019 Feb 1;74(2):425-431. doi: 10.1093/jac/dky439. PMID 30380060
- [Derived] Taboada M, Melnick D, Iaconis JP, Sun F, Zhong NS, File TM, Llorens L, Friedland HD, Wilson D. Ceftaroline fosamil versus ceftriaxone for the treatment of community-acquired pneumonia: individual patient data meta-analysis of randomized controlled trials. J Antimicrob Chemother. 2016 Apr;71(4):862-70. doi: 10.1093/jac/dkv415. Epub 2015 Dec 24. PMID 26702925
- [Derived] Zhong NS, Sun T, Zhuo C, D'Souza G, Lee SH, Lan NH, Chiang CH, Wilson D, Sun F, Iaconis J, Melnick D. Ceftaroline fosamil versus ceftriaxone for the treatment of Asian patients with community-acquired pneumonia: a randomised, controlled, double-blind, phase 3, non-inferiority with nested superiority trial. Lancet Infect Dis. 2015 Feb;15(2):161-71. doi: 10.1016/S1473-3099(14)71018-7. Epub 2014 Dec 22. PMID 25539586
- See also: D3720C00002 CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1374&filename=D3720C00002_Synopsis.pdf
- See also: Revised CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1374&filename=D3720C00002_Revised_CSP_1_(redacted).pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period was from 13 December 2011 to 26 April 2013
Pre-assignment Details: Enrolled patients (patients who gave informed consent) were screened for up to 24 hours to ensure eligibility before being randomized
Groups:
- Ceftaroline 600mg: Ceftaroline fosamil was administered in two consecutive 300-mg IV infusions over 30 minutes, every 12 hours (q12h)
- Ceftriaxone 2g: Ceftriaxone for Injection is supplied as 1 g/vial (2 vials for a 2 grams dose) and a 2 grams dose infused over 30 (±10) minutes q24h (±2h).
Period: Overall Study
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Started | 381 | 383
Completed | 332 | 317
Not Completed | 49 | 66
Not completed — Withdrawal by Subject | 27 | 33
Not completed — Lost to Follow-up | 10 | 20
Not completed — Death | 3 | 4
Not completed — Protocol Violation | 3 | 0
Not completed — Investigator Decision | 3 | 8
Not completed — Last follow-up visit not conducted | 2 | 0
Not completed — Lack of therapeutic response | 0 | 1
Not completed — Surgery | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects who were intended to receive study treatment and were of PORT risk class III and IV. There was one patient with PORT risk class II who was not included in baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g | Total
Number analyzed (Participants) | 381 | 382 | 763
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (14.70) [21 to 94] | 65.8 (13.86) [19 to 92] | 66.0 (14.28) [19 to 94]
Age, Customized [Number; unit: Participants]
  <65 years | 155 | 146 | 301
  >=65 years | 226 | 236 | 462
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 110 | 226
  Male | 265 | 272 | 537
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 381 | 382 | 763

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate for Ceftaroline Compared to That for Ceftriaxone at Test of Cure (TOC) in CE Population
Description: Cure:Total resolution of all signs and symptoms of pneumonia (ie,CABP), or improvement to such an extent that further antimicrobial therapy was not necessary Failure: Any of the following: •Persistence, incomplete clinical resolution, or worsening in signs and symptoms of CABP that required alternative antimicrobial therapy •Treatment-limiting AE leading to discontinuation of study drug therapy, when subject required alternative antimicrobial therapy to treat the pneumonia •Death wherein pneumonia (ie,CABP) was considered causative Indeterminate: Inability to determine an outcome
Time Frame: 7-20 days after last dose of study drug
Population: CE population: All patients in the MITT population who also meet the minimal disease criteria for CABP and for whom sufficient information regarding CABP is available to determine the patient's outcome (ie, the patient does not have an indeterminate outcome).
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 258 | 240
Participants
  Clinical Cure | 217 | 178
  Clinical Failure | 41 | 62
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; The primary objective of this study was to determine the noninferiority in the clinical cure rate for ceftaroline compared to that for ceftriaxone at TOC in the CE in adult subjects with CABP; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the observed difference in the primary outcome measure (clinical cure rate) between the ceftaroline group and the ceftriaxone group was calculated in CE Population at the TOC visit. Noninferiority was concluded if the lower limit of the 95% CI was higher than -10% in CE Population. If non-inferioirity was achieved then a test of superioirty was conducted whereby if lower limit of 95% CI for the difference was >0% superioirty was concluded; RD is Ceftaroline clinical cure rate minus Ceftriaxone clinical cure rate. The CI was calculated by Miettinen and Nurminen method without adjustment; Risk Difference (RD) = 9.9, 95% CI 2-sided [2.8 to 17.1] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments

2. Secondary Outcome: Clinical Response at End of Treatment (EOT) Visit in MITT Population
Time Frame: Last day of study drug administration
Population: All randomized subjects who were intended to receive study treatment and were of PORT risk class III and IV.
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 381 | 382
Participants
  Clinical Cure | 321 | 281
  Clinical Failure | 45 | 82
  Indeterminate | 15 | 19
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; Test type: Superiority or Other; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 10.7, 95% CI 2-sided [4.9 to 16.4] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments

3. Secondary Outcome: Clinical Response at End of Treatment (EOT) Visit in CE Population
Time Frame: Last day of study drug administration
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 258 | 240
Participants
  Clinical Cure | 222 | 186
  Clinical Failure | 36 | 54
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; Test type: Superiority or Other; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 8.5, 95% CI 2-sided [1.8 to 15.4] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments

4. Secondary Outcome: Clinical Response at the Test of Cure (TOC) Visit in MITT Population
Time Frame: 7-20 days after last day of study drug administration
Population: All randomized subjects who were intended to receive study treatment and were of PORT risk class III and IV.
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 381 | 382
Participants
  Clinical Cure | 305 | 256
  Clinical Failure | 53 | 91
  Indeterminate | 23 | 35
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; Test type: Superiority or Other; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 13.0, 95% CI 2-sided [6.8 to 19.2] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments. If lower limit of 95% CI for the risk difference was >0% superioirty was concluded in this population

5. Secondary Outcome: Clinical Response at the Test of Cure (TOC) Visit in mMITT Population
Time Frame: 7-20 days after last day of study drug administration
Population: mMITT population: All subjects in MITT population who meet the minimal disease criteria for CABP and who have at least one typical bacterial organism consistent with a CABP pathogen identified from an appropriate microbiological specimen (eg, blood, sputum, or pleural fluid).
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 80 | 96
Participants
  Clinical Cure | 68 | 67
  Clinical Failure | 9 | 21
  Indeterminate | 3 | 8
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; Test type: Superiority or Other; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 15.2, 95% CI 2-sided [2.7 to 27.1] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments

6. Secondary Outcome: Clinical Response at the Test of Cure (TOC) Visit in ME Population
Time Frame: 7-20 days after last day of study drug administration
Population: ME population: The ME population includes patients who meet criteria for both the CE and mMITT populations.
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 57 | 62
Participants
  Clinical Cure | 50 | 47
  Clinical Failure | 7 | 15
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; Test type: Superiority or Other; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 11.9, 95% CI 2-sided [-2.2 to 25.8] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments

7. Secondary Outcome: Clinical Response at Test of Cure (TOC) Visit by Pathogen in ME Population
Time Frame: 7-20 days after last dose of study drug
Population: ME population: includes patients who meet criteria for both the CE and mMITT populations. In fact, there were different pathogens isolated and we decided to focus on the 5 ones that occurred the most. Additionally please be informed that patients number will not match even if we present all 18 pathogens due to polymicrobial infections.
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 57 | 62
Participants
  Staphylococcus aureus | 4 | 4
  Clinical Cure - Staphylococcus aureus | 4 | 2
  Clinical Failure - Staphylococcus aureus | 0 | 2
  Streptococcus pneumoniae | 22 | 15
  Clinical Cure - Streptococcus pneumoniae | 19 | 13
  Clinical Failure - Streptococcus pneumoniae | 3 | 2
  Escherichia coli | 3 | 6
  Clinical Cure - Escherichia coli | 3 | 5
  Clinical Failure - Escherichia coli | 0 | 1
  Haemophilus influenzae | 12 | 7
  Clinical Cure - Haemophilus influenzae | 11 | 6
  Clinical Failure - Haemophilus influenzae | 1 | 1
  Klebsiella pneumoniae | 14 | 16
  Clinical Cure - Klebsiella pneumoniae | 11 | 12
  Clinical Failure - Klebsiella pneumoniae | 3 | 4

8. Secondary Outcome: Per-Pathogen Microbiological Response at Test of Cure (TOC) Visit by Pathogen in ME Population
Time Frame: 7-20 days after last dose of study drug
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 57 | 62
Participants
  Staphylococcus aureus | 4 | 4
  Favourable - Staphylococcus aureus | 4 | 2
  Unfavourable - Staphylococcus aureus | 0 | 2
  Streptococcus pneumoniae | 22 | 15
  Favourable - Streptococcus pneumoniae | 19 | 13
  Unfavourable - Streptococcus pneumoniae | 3 | 2
  Escherichia coli | 3 | 6
  Favourable - Escherichia coli | 3 | 5
  Unfavourable - Escherichia coli | 0 | 1
  Haemophilus influenzae | 12 | 7
  Favourable - Haemophilus influenzae | 11 | 6
  Unfavourable - Haemophilus influenzae | 1 | 1
  Klebsiella pneumoniae | 14 | 16
  Favourable - Klebsiella pneumoniae | 11 | 12
  Unfavourable - Klebsiella pneumoniae | 3 | 4

9. Secondary Outcome: Per-Patient Microbiological Response at Test of Cure (TOC) Visit in mMITT Population
Description: An outcome is considered as favourable if the per-pathogen response for that subject is either Eradication (An adequate source specimen demonstrates absence of the original baseline pathogen) or presumed eradication (An adequate source specimen was not available to culture and the patient was assessed as a clinical cure). Here, an adequate source specimen is defined as any sample that may yield the growth of a CABP pathogen eg, blood, respiratory specimens, or pleural fluid.
Time Frame: 7-20 days after last day of study drug administration
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 80 | 96
Participants
  Favourable | 68 | 67
  Unfavourable | 9 | 21
  Indeterminate | 3 | 8
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; Test type: Superiority or Other; RD is (Ceftaroline-Ceftriaxone) microbiologically favourable outcome rate. The CI was calculated by Miettinen and Nurminen method without adjustment; Risk Difference (RD) = 15.2, 95% CI 2-sided [2.7 to 27.1] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments

10. Secondary Outcome: Per-Patient Microbiological Response at Test of Cure (TOC) Visit in ME Population
Description: as for outcome 9
Time Frame: 7-20 days after last day of study drug administration
Population: ME population: The ME population includes patients who meet criteria for both the CE and mMITT populations.
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 57 | 62
Participants
  Favourable | 50 | 47
  Unfavourable | 7 | 15
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; Test type: Superiority or Other; [statistical method as in outcome 9, analysis 1]; Risk Difference (RD) = 11.9, 95% CI 2-sided [-2.2 to 25.8] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments

11. Secondary Outcome: Overall (Clinical and Radiographic) Success Rate at Test of Cure (TOC) Visit in MITT Population
Time Frame: 7-20 days after last day of study drug administration
Population: All randomized subjects who were intended to receive study treatment and were of PORT risk class III and IV.
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 381 | 382
Participants
  Success | 305 | 256
  Failure | 53 | 91
  Indeterminate | 23 | 35
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; Test type: Superiority or Other; RD is Ceftaroline minus Ceftriaxone overall success rate. The CI was calculated by Miettinen and Nurminen method without adjustment; Risk Difference (RD) = 13.0, 95% CI 2-sided [6.8 to 19.2] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments

12. Secondary Outcome: Overall (Clinical and Radiographic) Success Rate at Test of Cure (TOC) Visit in CE Population
Time Frame: 7-20 days after last dose of study drug
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 258 | 240
Participants
  Success | 217 | 178
  Failure | 41 | 62
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; Test type: Superiority or Other; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 9.9, 95% CI 2-sided [2.8 to 17.1] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments

13. Secondary Outcome: Clinical Relapse at the LFU Visit for Clinical Cure Patients at Test of Cure (TOC) Visit in MITT Population
Time Frame: 21-42 days after last day of study drug administration
Population: All randomized subjects who were intended to receive study treatment and were of PORT risk class III and IV. For this measure only patients who were cured at TOC could be assessed for relapse.
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 305 | 256
Participants
  Clinical relapse | 286 | 244
  No Clinical relapse | 7 | 5
  Indeterminate | 12 | 7
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; Test type: Superiority or Other; RD is Ceftaroline minus Ceftriaxone No-relapse rate. The CI was calculated by Miettinen and Nurminen method without adjustment; Risk Difference (RD) = 0.3, 95% CI 2-sided [-2.5 to 3.0] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments

14. Secondary Outcome: Clinical Relapse at the LFU Visit for Clinical Cure Patients at Test of Cure (TOC) Visit in CE Population
Time Frame: 21-42 days after last day of study drug administration
Population: CE population: All patients in the MITT population who also meet the minimal disease criteria for CABP and for whom sufficient information regarding CABP is available to determine the patient's outcome (ie, the patient does not have an indeterminate outcome). For this measure only patients who were cured at TOC could be assessed for relapse.
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 217 | 178
Participants
  Clinical relapse | 199 | 167
  No Clinical relapse | 6 | 3
  Indeterminate | 12 | 8
Statistical Analysis 1: Comparison: Ceftaroline 600mg vs Ceftriaxone 2g; Test type: Superiority or Other; [statistical method as in outcome 13, analysis 1]; Risk Difference (RD) = 1.1, 95% CI 2-sided [-2.4 to 4.5] — CI for risk difference was estimated by 95% Miettinen and Nurminen CI without adjustments

15. Secondary Outcome: Microbiological Re-infection/Recurrence at LFU Visit in mMITT Population
Time Frame: 21-42 days after last dose of study drug
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 80 | 96
Participants
  Super-Infection | 0 | 2
  Favourable response at TOC | 68 | 67
  No Re-Infection Or Recurrance | 68 | 66
  Re-Infection Or Recurrance | 0 | 1

16. Secondary Outcome: Microbiological Re-infection/Recurrence at LFU Visit in ME Population
Time Frame: 21-42 days after last dose of study drug
Population: ME population: The ME population includes patients who meet criteria for both the CE and mMITT populations
Measure: Number; unit: Participants
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Number analyzed (Participants) | 57 | 62
Participants
  Super-Infection | 0 | 1
  Favourable response at TOC | 50 | 47
  No Re-Infection Or Recurrance | 50 | 46
  Re-Infection Or Recurrance | 0 | 1

ADVERSE EVENTS:
Time Frame: first dose, throughout the treatment period, and up to the TOC visit
Description: All adverse events with an onset date between the date of first dose and test of cure (TOC) or 20 days following the EOT in absence of TOC and all serious adverse events with an onset date between the date of first dose and test of cure (TOC) or 30 days following the EOT in absence of TOC.
Arm/Group | Ceftaroline 600mg | Ceftriaxone 2g
Serious Adverse Events (participants affected / at risk) | 30/381 | 29/383
Other Adverse Events (participants affected / at risk) | 24/381 | 13/383
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline 600mg (N=381) | Ceftriaxone 2g (N=383)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
ASPERGILLOSIS (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 (0) | 2 (2)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1)
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
GOUT (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COMA (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS (Vascular disorders) | 1 (1) | 1 (1)
HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSIVE EMERGENCY (Vascular disorders) | 1 (1) | 0 (0)
SHOCK (Vascular disorders) | 0 (0) | 1 (1)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1) | 0 (0)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline 600mg (N=381) | Ceftriaxone 2g (N=383)
DIARRHOEA (Gastrointestinal disorders) | 24 (24) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other